CLINICAL TRIAL: NCT02583516
Title: A Randomized Phase II Study of Vemurafenib Plus Cobimetinib Continuous Versus Intermittent, in Previously Untreated BRAFV600- Mutation Positive Patients With Unresectable Locally Advanced or Metastatic Melanoma
Brief Title: Clinical Trial to Evaluate the Efficacy of Vemurafenib in Combination With Cobimetinib (Continuous and Intermittent) in BRAFV600-mutation Positive Patients With Unresectable Locally Advanced or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: Roche Farma, S.A (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-01-15; 2014-005277-36 (EudraCT Number)
Record Dates: First submitted 2015-10-08; First posted 2015-10-22 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Continuous Administration (Experimental): 960 mg of vemurafenib po, bid, days 1 to 28 and 60 mg of cobimetinib po, od, days 1 to 21, for each 28-days' cycle.
  Interventions: Drug: vemurafenib and cobimetinib
- B - Intermittent Administration (Experimental): 960 mg of vemurafenib po, bid, days 1 to 28 and 60 mg of cobimetinib po, od, days 1 to 21, for each 28-days' cycle, during 12 weeks. After that period, patients will be treated with both drugs at the same doses indicated previously, but with an intermittent pattern: vemurafenib days 1 to 28 followed by 14 days off (4 weeks on and 2 weeks off) and cobimetinib days 1 to 21 followed by 21 days off (3 weeks on and 3 weeks off)
  Interventions: Drug: vemurafenib and cobimetinib

INTERVENTIONS:
Drug: vemurafenib and cobimetinib — Comparison between different treatment regimens

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two different schedules of administration of vemurafenib in combination with cobimetinib (continuous and intermittent) in previously untreated BRAFV600- mutation positive patients with unresectable locally advanced or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

Disease-Specific Inclusion Criteria:

1. Patients with histologically confirmed melanoma, either unresectable stage IIIc or stage IV metastatic melanoma.
2. Patients must be naïve to treatment for locally advanced unresectable or metastatic disease.
3. Documentation of BRAFV600 mutation-positive status in melanoma tumor tissue.
4. Measurable disease per RECIST v1.1.
5. ECOG performance status of 0 or 1.
6. Additionally, patients to be included in the biomarker sub- study should meet the following criteria:

   * Consent to provide archival tissue for biomarker analyses.
   * Consent to undergo tumor biopsies.

   General Inclusion Criteria:
7. Male or female patient aged major or equal 18 years.
8. Able to participate and willing to give written informed.
9. Life expectancy mayor o igual 12 weeks.
10. Adequate hematologic and end organ function, within 14 days prior to first dose of study drug treatment:

    * ANC major or equal 1.5 × 109/L.
    * Platelet count major or equal 100 × 109/L.
    * Hemoglobin major or equal 9 g/dL.
    * Albumin major or equal 2.5 g/dL.
    * Bilirubin minor or equal 1.5 × the upper limit of normal (ULN).
    * AST, ALT, and alkaline phosphatase minor or equal 3 × ULN, with the following exceptions:
    * Patients with documented liver metastases: AST and/or ALT minor or equal 5 × ULN.
    * Patients with documented liver or bone metastases alkaline phosphatase minor o equal 5 × ULN.
    * Serum creatinine minor o equal 1.5 × ULN or CrCl major or equal 40 mL/min on the basis of measured CrCl from a 24- hour urine collection.
11. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to always use 2 effective forms of contraception during the course of this study and for at least 6 months after completion of study therapy.
12. Negative serum pregnancy test within 10 days prior to commencement of dosing in women of childbearing potential.
13. Absence of any psychological, familial, sociological, or geographical condition that potentially hampers compliance with the study protocol and follow-up after treatment discontinuation schedule.

Exclusion Criteria:

Cancer-Related Exclusion Criteria:

1. History of prior RAF or MEK pathway inhibitor treatment.
2. Palliative radiotherapy within 14 days prior to the first dose of study treatment.
3. Major surgery or traumatic injury within 14 days prior to first dose of study treatment.
4. Active malignancy other than melanoma that could potentially interfere with the interpretation of efficacy measures. Patients with a previous malignancy within the past 3 years are excluded except for patients with resected BCC or SCC of the skin, melanoma in-situ, carcinoma in-situ of the cervix, and carcinoma in-situ of the breast. History of isolated elevation in prostate-specific antigen in the absence of radiographic evidence of metastatic prostate cancer is allowed.

   Exclusion Criteria Based on Ocular Function:
5. History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, retinal vein occlusion (RVO), or neovascular macular degeneration.

   The risk factors for RVO are listed below. Patients will be excluded if they have the following conditions:
   * Uncontrolled glaucoma with intra-ocular pressures > 21 mmHg.
   * Serum cholesterol major or equal Grade 2.
   * Hypertriglyceridemia major or equal Grade 2.
   * Hyperglycemia (fasting) major or equal Grade 2.

   Exclusion Criteria Based on Cardiac Function:
6. History of clinically significant cardiac dysfunction, including the following:

   * Current unstable angina.
   * Symptomatic congestive heart failure of New York Heart Association class 2 or higher.
   * History of congenital long QT syndrome or mean (average of triplicate measurements) QTcF > 450 msec at baseline or uncorrectable abnormalities in serum electrolytes (sodium, potassium, calcium, magnesium, phosphorus). If not automated, calculation of QTcF must be done through the following formula: QTcF = (QT interval in ms) / [(60 / heart rate in bpm) )^(1/3)]
   * Uncontrolled hypertension major or equal Grade 2 (patients with a history hypertension controlled with anti-hypertensives to minor or equal Grade 1 are eligible).
   * Left ventricular ejection fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%.

   Exclusion Criteria Based on Central Nervous System Function:
7. Patients with active CNS lesions (including melanomatous meningitis) are excluded. However, patients are eligible if:

   * All known CNS lesions have been treated with stereotactic therapy or surgery, AND
   * There has been no evidence of clinical and radiographic disease progression in the CNS for major or equal 3 weeks after radiotherapy or surgery.

   Whole brain radiotherapy is not allowed, with the exception of patients who have had definitive resection or stereotactic therapy of all radiologically detectable parenchymal brain lesions.

   General Exclusion Criteria:
8. Current severe, uncontrolled systemic disease.
9. History of malabsorption or other condition that would interfere with absorption of study drugs.
10. Pregnant or lactating.
11. Unwillingness or inability to comply with study and follow- up procedures.
12. The following foods/supplements are prohibited at least 7 days prior to initiation of and during study treatment:

    * St. Johns wort or hyperforin (potent cytochrome P450 CYP3A4 enzyme inducer).
    * Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Through study completion, up to 42 months

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, up to 42 months
Progression Free Survival (PFS) at one and two years | At one and two years
Overall Survival (OS) at one and two years | At one and two years
Adverse Events (AE) occurrence | Through study completion, up to 42 months
Serious Adverse Events (SAE) occurrence | Through study completion, up to 42 months
Adverse Events of Special Interest (AESI) occurrence | Through study completion, up to 42 months

OTHER OUTCOMES:
BRAF mutation determination (Translational sub-study) | Through study completion, up to 42 months
  Analysis of prognostic and predictive value of BRAF mutation in cell-free DNA (cfDNA) samples, and its role in disease evolution monitoring.
Analysis of resistance mechanisms to the combination of vemurafenib and cobimetinib (Translational sub-study) | Through study completion, up to 42 months
  Non-invasive monitorization of resistance mechanisms, through selected gene expression cuantification from blood mRNA.
Analysis of disease's resistance mechanisms (Translational sub-study) | Through study completion, up to 42 months
  Determination of resistance mechanisms in secuential biopsies of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio López-Martín, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre; Alfonso Berrocal, MD, PhD, Principal Investigator — Hospital General Universitario de Valencia
Locations (18):
- Spain (18):
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Álvaro Cunqueiro (Complejo Hospitalario Universitario de Vigo), Vigo
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garbe C, Peris K, Hauschild A, Saiag P, Middleton M, Spatz A, Grob JJ, Malvehy J, Newton-Bishop J, Stratigos A, Pehamberger H, Eggermont A. Diagnosis and treatment of melanoma: European consensus-based interdisciplinary guideline. Eur J Cancer. 2010 Jan;46(2):270-83. doi: 10.1016/j.ejca.2009.10.032. Epub 2009 Dec 1. PMID 19959353
- [Background] Balch CM, Gershenwald JE, Soong SJ, Thompson JF, Atkins MB, Byrd DR, Buzaid AC, Cochran AJ, Coit DG, Ding S, Eggermont AM, Flaherty KT, Gimotty PA, Kirkwood JM, McMasters KM, Mihm MC Jr, Morton DL, Ross MI, Sober AJ, Sondak VK. Final version of 2009 AJCC melanoma staging and classification. J Clin Oncol. 2009 Dec 20;27(36):6199-206. doi: 10.1200/JCO.2009.23.4799. Epub 2009 Nov 16. PMID 19917835
- [Background] Avril MF, Aamdal S, Grob JJ, Hauschild A, Mohr P, Bonerandi JJ, Weichenthal M, Neuber K, Bieber T, Gilde K, Guillem Porta V, Fra J, Bonneterre J, Saiag P, Kamanabrou D, Pehamberger H, Sufliarsky J, Gonzalez Larriba JL, Scherrer A, Menu Y. Fotemustine compared with dacarbazine in patients with disseminated malignant melanoma: a phase III study. J Clin Oncol. 2004 Mar 15;22(6):1118-25. doi: 10.1200/JCO.2004.04.165. PMID 15020614
- [Background] Bedikian AY, Millward M, Pehamberger H, Conry R, Gore M, Trefzer U, Pavlick AC, DeConti R, Hersh EM, Hersey P, Kirkwood JM, Haluska FG; Oblimersen Melanoma Study Group. Bcl-2 antisense (oblimersen sodium) plus dacarbazine in patients with advanced melanoma: the Oblimersen Melanoma Study Group. J Clin Oncol. 2006 Oct 10;24(29):4738-45. doi: 10.1200/JCO.2006.06.0483. Epub 2006 Sep 11. PMID 16966688
- [Background] Middleton MR, Grob JJ, Aaronson N, Fierlbeck G, Tilgen W, Seiter S, Gore M, Aamdal S, Cebon J, Coates A, Dreno B, Henz M, Schadendorf D, Kapp A, Weiss J, Fraass U, Statkevich P, Muller M, Thatcher N. Randomized phase III study of temozolomide versus dacarbazine in the treatment of patients with advanced metastatic malignant melanoma. J Clin Oncol. 2000 Jan;18(1):158-66. doi: 10.1200/JCO.2000.18.1.158. PMID 10623706
- [Background] Eggermont AM, Schadendorf D. Melanoma and immunotherapy. Hematol Oncol Clin North Am. 2009 Jun;23(3):547-64, ix-x. doi: 10.1016/j.hoc.2009.03.009. PMID 19464602
- [Background] Hauschild A, Agarwala SS, Trefzer U, Hogg D, Robert C, Hersey P, Eggermont A, Grabbe S, Gonzalez R, Gille J, Peschel C, Schadendorf D, Garbe C, O'Day S, Daud A, White JM, Xia C, Patel K, Kirkwood JM, Keilholz U. Results of a phase III, randomized, placebo-controlled study of sorafenib in combination with carboplatin and paclitaxel as second-line treatment in patients with unresectable stage III or stage IV melanoma. J Clin Oncol. 2009 Jun 10;27(17):2823-30. doi: 10.1200/JCO.2007.15.7636. Epub 2009 Apr 6. PMID 19349552
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Robert C, Thomas L, Bondarenko I, O'Day S, Weber J, Garbe C, Lebbe C, Baurain JF, Testori A, Grob JJ, Davidson N, Richards J, Maio M, Hauschild A, Miller WH Jr, Gascon P, Lotem M, Harmankaya K, Ibrahim R, Francis S, Chen TT, Humphrey R, Hoos A, Wolchok JD. Ipilimumab plus dacarbazine for previously untreated metastatic melanoma. N Engl J Med. 2011 Jun 30;364(26):2517-26. doi: 10.1056/NEJMoa1104621. Epub 2011 Jun 5. PMID 21639810
- [Background] Curtin JA, Fridlyand J, Kageshita T, Patel HN, Busam KJ, Kutzner H, Cho KH, Aiba S, Brocker EB, LeBoit PE, Pinkel D, Bastian BC. Distinct sets of genetic alterations in melanoma. N Engl J Med. 2005 Nov 17;353(20):2135-47. doi: 10.1056/NEJMoa050092. PMID 16291983
- [Background] Davies H, Bignell GR, Cox C, Stephens P, Edkins S, Clegg S, Teague J, Woffendin H, Garnett MJ, Bottomley W, Davis N, Dicks E, Ewing R, Floyd Y, Gray K, Hall S, Hawes R, Hughes J, Kosmidou V, Menzies A, Mould C, Parker A, Stevens C, Watt S, Hooper S, Wilson R, Jayatilake H, Gusterson BA, Cooper C, Shipley J, Hargrave D, Pritchard-Jones K, Maitland N, Chenevix-Trench G, Riggins GJ, Bigner DD, Palmieri G, Cossu A, Flanagan A, Nicholson A, Ho JW, Leung SY, Yuen ST, Weber BL, Seigler HF, Darrow TL, Paterson H, Marais R, Marshall CJ, Wooster R, Stratton MR, Futreal PA. Mutations of the BRAF gene in human cancer. Nature. 2002 Jun 27;417(6892):949-54. doi: 10.1038/nature00766. Epub 2002 Jun 9. PMID 12068308
- [Background] Gray-Schopfer V, Wellbrock C, Marais R. Melanoma biology and new targeted therapy. Nature. 2007 Feb 22;445(7130):851-7. doi: 10.1038/nature05661. PMID 17314971
- [Background] Bollag G, Hirth P, Tsai J, Zhang J, Ibrahim PN, Cho H, Spevak W, Zhang C, Zhang Y, Habets G, Burton EA, Wong B, Tsang G, West BL, Powell B, Shellooe R, Marimuthu A, Nguyen H, Zhang KY, Artis DR, Schlessinger J, Su F, Higgins B, Iyer R, D'Andrea K, Koehler A, Stumm M, Lin PS, Lee RJ, Grippo J, Puzanov I, Kim KB, Ribas A, McArthur GA, Sosman JA, Chapman PB, Flaherty KT, Xu X, Nathanson KL, Nolop K. Clinical efficacy of a RAF inhibitor needs broad target blockade in BRAF-mutant melanoma. Nature. 2010 Sep 30;467(7315):596-9. doi: 10.1038/nature09454. PMID 20823850
- [Background] Flaherty KT, Puzanov I, Kim KB, Ribas A, McArthur GA, Sosman JA, O'Dwyer PJ, Lee RJ, Grippo JF, Nolop K, Chapman PB. Inhibition of mutated, activated BRAF in metastatic melanoma. N Engl J Med. 2010 Aug 26;363(9):809-19. doi: 10.1056/NEJMoa1002011. PMID 20818844
- [Background] Joseph EW, Pratilas CA, Poulikakos PI, Tadi M, Wang W, Taylor BS, Halilovic E, Persaud Y, Xing F, Viale A, Tsai J, Chapman PB, Bollag G, Solit DB, Rosen N. The RAF inhibitor PLX4032 inhibits ERK signaling and tumor cell proliferation in a V600E BRAF-selective manner. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14903-8. doi: 10.1073/pnas.1008990107. Epub 2010 Jul 28. PMID 20668238
- [Background] Tsai J, Lee JT, Wang W, Zhang J, Cho H, Mamo S, Bremer R, Gillette S, Kong J, Haass NK, Sproesser K, Li L, Smalley KS, Fong D, Zhu YL, Marimuthu A, Nguyen H, Lam B, Liu J, Cheung I, Rice J, Suzuki Y, Luu C, Settachatgul C, Shellooe R, Cantwell J, Kim SH, Schlessinger J, Zhang KY, West BL, Powell B, Habets G, Zhang C, Ibrahim PN, Hirth P, Artis DR, Herlyn M, Bollag G. Discovery of a selective inhibitor of oncogenic B-Raf kinase with potent antimelanoma activity. Proc Natl Acad Sci U S A. 2008 Feb 26;105(8):3041-6. doi: 10.1073/pnas.0711741105. Epub 2008 Feb 19. PMID 18287029
- [Background] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808
- [Background] Johannessen CM, Boehm JS, Kim SY, Thomas SR, Wardwell L, Johnson LA, Emery CM, Stransky N, Cogdill AP, Barretina J, Caponigro G, Hieronymus H, Murray RR, Salehi-Ashtiani K, Hill DE, Vidal M, Zhao JJ, Yang X, Alkan O, Kim S, Harris JL, Wilson CJ, Myer VE, Finan PM, Root DE, Roberts TM, Golub T, Flaherty KT, Dummer R, Weber BL, Sellers WR, Schlegel R, Wargo JA, Hahn WC, Garraway LA. COT drives resistance to RAF inhibition through MAP kinase pathway reactivation. Nature. 2010 Dec 16;468(7326):968-72. doi: 10.1038/nature09627. Epub 2010 Nov 24. PMID 21107320
- [Background] Nazarian R, Shi H, Wang Q, Kong X, Koya RC, Lee H, Chen Z, Lee MK, Attar N, Sazegar H, Chodon T, Nelson SF, McArthur G, Sosman JA, Ribas A, Lo RS. Melanomas acquire resistance to B-RAF(V600E) inhibition by RTK or N-RAS upregulation. Nature. 2010 Dec 16;468(7326):973-7. doi: 10.1038/nature09626. Epub 2010 Nov 24. PMID 21107323
- [Background] Poulikakos PI, Persaud Y, Janakiraman M, Kong X, Ng C, Moriceau G, Shi H, Atefi M, Titz B, Gabay MT, Salton M, Dahlman KB, Tadi M, Wargo JA, Flaherty KT, Kelley MC, Misteli T, Chapman PB, Sosman JA, Graeber TG, Ribas A, Lo RS, Rosen N, Solit DB. RAF inhibitor resistance is mediated by dimerization of aberrantly spliced BRAF(V600E). Nature. 2011 Nov 23;480(7377):387-90. doi: 10.1038/nature10662. PMID 22113612
- [Background] Shi H, Moriceau G, Kong X, Lee MK, Lee H, Koya RC, Ng C, Chodon T, Scolyer RA, Dahlman KB, Sosman JA, Kefford RF, Long GV, Nelson SF, Ribas A, Lo RS. Melanoma whole-exome sequencing identifies (V600E)B-RAF amplification-mediated acquired B-RAF inhibitor resistance. Nat Commun. 2012 Mar 6;3:724. doi: 10.1038/ncomms1727. PMID 22395615
- [Background] Su F, Bradley WD, Wang Q, Yang H, Xu L, Higgins B, Kolinsky K, Packman K, Kim MJ, Trunzer K, Lee RJ, Schostack K, Carter J, Albert T, Germer S, Rosinski J, Martin M, Simcox ME, Lestini B, Heimbrook D, Bollag G. Resistance to selective BRAF inhibition can be mediated by modest upstream pathway activation. Cancer Res. 2012 Feb 15;72(4):969-78. doi: 10.1158/0008-5472.CAN-11-1875. Epub 2011 Dec 28. PMID 22205714
- [Background] Villanueva J, Vultur A, Lee JT, Somasundaram R, Fukunaga-Kalabis M, Cipolla AK, Wubbenhorst B, Xu X, Gimotty PA, Kee D, Santiago-Walker AE, Letrero R, D'Andrea K, Pushparajan A, Hayden JE, Brown KD, Laquerre S, McArthur GA, Sosman JA, Nathanson KL, Herlyn M. Acquired resistance to BRAF inhibitors mediated by a RAF kinase switch in melanoma can be overcome by cotargeting MEK and IGF-1R/PI3K. Cancer Cell. 2010 Dec 14;18(6):683-95. doi: 10.1016/j.ccr.2010.11.023. PMID 21156289
- [Background] Wagle N, Emery C, Berger MF, Davis MJ, Sawyer A, Pochanard P, Kehoe SM, Johannessen CM, Macconaill LE, Hahn WC, Meyerson M, Garraway LA. Dissecting therapeutic resistance to RAF inhibition in melanoma by tumor genomic profiling. J Clin Oncol. 2011 Aug 1;29(22):3085-96. doi: 10.1200/JCO.2010.33.2312. Epub 2011 Mar 7. PMID 21383288
- [Background] Atefi M, von Euw E, Attar N, Ng C, Chu C, Guo D, Nazarian R, Chmielowski B, Glaspy JA, Comin-Anduix B, Mischel PS, Lo RS, Ribas A. Reversing melanoma cross-resistance to BRAF and MEK inhibitors by co-targeting the AKT/mTOR pathway. PLoS One. 2011;6(12):e28973. doi: 10.1371/journal.pone.0028973. Epub 2011 Dec 14. PMID 22194965
- [Background] Paraiso KH, Fedorenko IV, Cantini LP, Munko AC, Hall M, Sondak VK, Messina JL, Flaherty KT, Smalley KS. Recovery of phospho-ERK activity allows melanoma cells to escape from BRAF inhibitor therapy. Br J Cancer. 2010 Jun 8;102(12):1724-30. doi: 10.1038/sj.bjc.6605714. PMID 20531415
- [Background] Ribas A, Gonzalez R, Pavlick A, Hamid O, Gajewski TF, Daud A, Flaherty L, Logan T, Chmielowski B, Lewis K, Kee D, Boasberg P, Yin M, Chan I, Musib L, Choong N, Puzanov I, McArthur GA. Combination of vemurafenib and cobimetinib in patients with advanced BRAF(V600)-mutated melanoma: a phase 1b study. Lancet Oncol. 2014 Aug;15(9):954-65. doi: 10.1016/S1470-2045(14)70301-8. Epub 2014 Jul 15. PMID 25037139
- [Background] Larkin J, Ascierto PA, Dreno B, Atkinson V, Liszkay G, Maio M, Mandala M, Demidov L, Stroyakovskiy D, Thomas L, de la Cruz-Merino L, Dutriaux C, Garbe C, Sovak MA, Chang I, Choong N, Hack SP, McArthur GA, Ribas A. Combined vemurafenib and cobimetinib in BRAF-mutated melanoma. N Engl J Med. 2014 Nov 13;371(20):1867-76. doi: 10.1056/NEJMoa1408868. Epub 2014 Sep 29. PMID 25265494
- [Background] Das Thakur M, Stuart DD. The evolution of melanoma resistance reveals therapeutic opportunities. Cancer Res. 2013 Oct 15;73(20):6106-10. doi: 10.1158/0008-5472.CAN-13-1633. Epub 2013 Oct 4. PMID 24097822
- [Background] Callahan MK, Rampal R, Harding JJ, Klimek VM, Chung YR, Merghoub T, Wolchok JD, Solit DB, Rosen N, Abdel-Wahab O, Levine RL, Chapman PB. Progression of RAS-mutant leukemia during RAF inhibitor treatment. N Engl J Med. 2012 Dec 13;367(24):2316-21. doi: 10.1056/NEJMoa1208958. Epub 2012 Nov 7. PMID 23134356
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Derived] Gonzalez-Cao M, Mayo de Las Casas C, Oramas J, Berciano-Guerrero MA, de la Cruz L, Cerezuela P, Arance A, Munoz-Couselo E, Espinosa E, Puertolas T, Diaz Beveridge R, Ochenduszko S, Villanueva MJ, Basterretxea L, Bellido L, Rodriguez D, Campos B, Montagut C, Drozdowskyj A, Molina MA, Lopez-Martin JA, Berrocal A. Intermittent BRAF inhibition in advanced BRAF mutated melanoma results of a phase II randomized trial. Nat Commun. 2021 Dec 1;12(1):7008. doi: 10.1038/s41467-021-26572-6. PMID 34853302
- See also: Spanish Multidisciplinary Melanoma Group Web — http://www.groupgem.org/